CLINICAL TRIAL: NCT02666755
Title: Novel Detection System for Detecting Epidermal Growth Factor Receptor Mutation in Plasma in Non-small Cell Lung Cancer
Brief Title: Novel Detection System for Lung Cancer Curative Effect Monitoring
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Jian Zhang (Other)
Responsible Party: Sponsor-Investigator, Jian Zhang, director of Respiration Department, Air Force Military Medical University, China
Organization: Air Force Military Medical University, China (Other)
Other Study IDs: 15229491635
Record Dates: First submitted 2016-01-19; First posted 2016-01-28 (Estimated); Last update posted 2016-01-29 (Estimated); Status verified 2016-01

CONDITIONS: Lung Neoplasms
Keywords: Lung Neoplasms digital polymerase chain reaction
MeSH Terms: conditions — Lung Neoplasms

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Each specimen was collected into one 10mL EDTA-containing vacutainer and was spun into plasma within 4 hours of collection. cfDNA was extracted from 2 mL of plasma, and the final DNA eluent was frozen at- 20℃ until genotyping
Oversight: Data Monitoring Committee: Yes

SUMMARY:
The purpose of this study is to investigate the sensitivity，specificity and concordance rate of EGFR testing results in plasma in comparison of results in matched tumor tissues tested by amplification refractory mutation system(ARMS). Moreover, the investigators correlate our findings in plasma with survival of advanced patients.

DETAILED DESCRIPTION:
Non-small cell lung cancer (NSCLC), accounting for 80% of all lung cancers, is a leading cause of cancer deaths worldwide. Inhibition of epidermal growth factor receptor (EGFR) kinase activity by EGFR tyrosine kinase inhibitors, such as gefitinib and erlotinib, can result in improved response and prolonged progression-free survival (PFS) in selected non-small cell lung cancer (NSCLC) patients harboring sensitizing EGFR mutations, especially the exon 19del and exon 21（L858R） mutations. Unfortunately, about 50%-60% patients who accept EGFR tyrosine kinase inhibitors with sensitizing mutations will receive resistance mutations, the T790M resistance is a target of active pharmaceutical development. So EGFR mutation testing is a step in identifying the right patients for EGFR tyrosine kinase inhibitors treatment. Now tissue samples and tumor cytologic samples are accepted as appropriate sample types for EGFR mutation detection, but these samples are not always available on or after diagnosis, and, even when available, they may be of insufficient quality or quantity for mutation testing. Noninvasive techniques for tumor genotyping may be needed to fully realize, such as plasma sample. Cell-free DNA (cf-DNA) in plasma is a kind of fresh and realtime sample, and has been shown to be promising for the detection of sensitizing EGFR mutations even the resistance mutation（T790M). However, a challenge was also raised about how to detect the low abundance of mutant alleles in plasma. In our study Droplet Digital polymerase chain reaction and Realtime polymerase chain reaction will be used to assess the EGFR mutation in plasma DNA samples from patients with advanced NSCLC before and after EGFR tyrosine kinase inhibitors therapy.

ELIGIBILITY:
Inclusion Criteria:

1. Aged 18-85 years old;
2. The diagnosis of lung cancer by pathological examination;
3. At least one specific measurable lung cancer lesions (according to RECIST criteria, application of spiral CT, the lesion diameter 10 mm or higher);
4. People understand and are willing to accept the study, and sign the informed consent

Exclusion Criteria:

1. With severe hemorrhagic disease;
2. Compliance is poor, can't cooperate with the visitor.

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: patients diagnosed with NSCLC
Sampling Method: Probability Sample
Enrollment: 160 (Estimated)
Dates: Start 2016-01; Primary Completion 2018-01 (Estimated); Study Completion 2018-04 (Estimated)

PRIMARY OUTCOMES:
sensitivity | 2 years
  comparing with results in tissues, tne investigators can get the sensitivity of results in plasma for Epidermal Growth Factor Receptor mutation in Non-small cell lung cancer.

SECONDARY OUTCOMES:
specificity | 2 years
  comparing with results in tissues, the investigators can get the specificity of results in plasma for Epidermal Growth Factor Receptor mutation in Non-small cell lung cancer.

CONTACTS AND LOCATIONS:
Overall Officials: Jian Zhang, Doctor, Study Director — Xijing Hospital

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Zhu G, Ye X, Dong Z, Lu YC, Sun Y, Liu Y, McCormack R, Gu Y, Liu X. Highly Sensitive Droplet Digital PCR Method for Detection of EGFR-Activating Mutations in Plasma Cell-Free DNA from Patients with Advanced Non-Small Cell Lung Cancer. J Mol Diagn. 2015 May;17(3):265-72. doi: 10.1016/j.jmoldx.2015.01.004. Epub 2015 Mar 11. PMID 25769900
- [Background] Jemal A, Bray F, Center MM, Ferlay J, Ward E, Forman D. Global cancer statistics. CA Cancer J Clin. 2011 Mar-Apr;61(2):69-90. doi: 10.3322/caac.20107. Epub 2011 Feb 4. PMID 21296855
- [Background] Mok TS, Wu YL, Thongprasert S, Yang CH, Chu DT, Saijo N, Sunpaweravong P, Han B, Margono B, Ichinose Y, Nishiwaki Y, Ohe Y, Yang JJ, Chewaskulyong B, Jiang H, Duffield EL, Watkins CL, Armour AA, Fukuoka M. Gefitinib or carboplatin-paclitaxel in pulmonary adenocarcinoma. N Engl J Med. 2009 Sep 3;361(10):947-57. doi: 10.1056/NEJMoa0810699. Epub 2009 Aug 19. PMID 19692680
- [Background] Zhou C, Wu YL, Chen G, Feng J, Liu XQ, Wang C, Zhang S, Wang J, Zhou S, Ren S, Lu S, Zhang L, Hu C, Hu C, Luo Y, Chen L, Ye M, Huang J, Zhi X, Zhang Y, Xiu Q, Ma J, Zhang L, You C. Erlotinib versus chemotherapy as first-line treatment for patients with advanced EGFR mutation-positive non-small-cell lung cancer (OPTIMAL, CTONG-0802): a multicentre, open-label, randomised, phase 3 study. Lancet Oncol. 2011 Aug;12(8):735-42. doi: 10.1016/S1470-2045(11)70184-X. Epub 2011 Jul 23. PMID 21783417
- [Result] Yu M, Bardia A, Wittner BS, Stott SL, Smas ME, Ting DT, Isakoff SJ, Ciciliano JC, Wells MN, Shah AM, Concannon KF, Donaldson MC, Sequist LV, Brachtel E, Sgroi D, Baselga J, Ramaswamy S, Toner M, Haber DA, Maheswaran S. Circulating breast tumor cells exhibit dynamic changes in epithelial and mesenchymal composition. Science. 2013 Feb 1;339(6119):580-4. doi: 10.1126/science.1228522. PMID 23372014